CLINICAL TRIAL: NCT04852094
Title: Family-centered Round in Neonatal Units : Process Development and Implementation Using the Intervention Mapping
Brief Title: Family-centered Round in Neonatology
Acronym: VINCI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: VINCI
Record Dates: First submitted 2021-04-11; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Prematurity
Keywords: Newborn; Preterm; medical round; family-centered care; NICU
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents: parents of hospitalized children, speaking and understanding enough French, not presenting psychiatric disorders, voluntary to participate in focus groups
  Interventions: Other: Qualitative focus group
- Professionals: Nurses, assistant nurses, psychologist, physiotherapist, physicians, residents and fellows
  Interventions: Other: Qualitative focus group

INTERVENTIONS:
Other: Qualitative focus group — A qualitative focus group is performed with staff members and parents of hospitalised newborns in a NICU during Family-centered rounds management. The transcribed interviews are analyzed with qualitative content analysis in order to illuminate the experience, feelings and thoughts arisen among the staff members and the parents.

SUMMARY:
The family-centered care is based on dignity and respect, information sharing, collaboration and participation in care and decision-making. In a neonatal unit, the medical round by the attending physician is an important moment for shairing information with the medical and nursing staff and for the decision making process. In France, parents are rarely actively involved in the medical round. The aim of this study is to plan the implantation of the Family-centered round in a neonatal department using the 6 steps of the "Intervention mapping": 1/needs assessment; 2/ performance and change objectives; 3/ theory-based framework; Curriculum development; 5- adoption and implementation; 6- evaluation and dissemination

ELIGIBILITY:
Parents Group:

Inclusion Criteria:

* French speaking
* voluntary to participate
* parents of an hospitalized newborn

Exclusion Criteria:

* not fluent in French speaking
* mental health problems

Professional group:

* any staff member
* voluntary to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents group: age, parity, education and income level Staff group: age, gender, years of experience in the NICU, profession
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Experience of participating to a Family-Centered Care (FCR) | 1 day during the last week of their newborn 'hospitalisation
  Qualitative focus group interview performed at one occasion where the parent describes the experience of the FCR

SECONDARY OUTCOMES:
Experience of staff members in participating to a (FCR) | 1 day after 3 months of FCR experience
  Qualitative focus group interview performed at one occasion where the staff members describes the experience of the FCR

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Sizun, Principal Investigator — University Hospital, Brest
Locations (1):
- CHRU de Brest, Brest, France